CLINICAL TRIAL: NCT04612504
Title: An Open-label Phase I Study to Evaluate the Safety, Tolerability and Efficacy of SynOV1.1 Recombinant Oncolytic Adenovirus Injection as Monotherapy in Participants With Locally Advanced or Metastatic Solid Tumors
Brief Title: SynOV1.1 Intratumoral Injection Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Syngentech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Syngentech-SynOV1.1-101
Record Dates: First submitted 2020-10-16; First posted 2020-11-03 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SynOV1.1 Injection (Experimental)
  Interventions: Biological: SynOV1.1

INTERVENTIONS:
Biological: SynOV1.1 — SynOV1.1 will be administered intratumorally.

SUMMARY:
This is a Phase I, open-label, multicenter study to characterize safety and tolerability, evaluate biodistribution, biological effects and immunogenicity, and evaluate the preliminary clinical efficacy of SynOV1.1 in participants with AFP positive solid tumors.

DETAILED DESCRIPTION:
Part 1 ( single dose escalation) is designed to determine the pharmacodynamics of SynOV1.1 as well as type and severity of toxicity based on safety and tolerability assessments. 3 dose level (3 × 10^11 Vp, 1 × 10^12 Vp, 3 × 10^12 Vp) will be evaluated.

Part 2 (multiple dose escalation) is designed to determine the pharmacodynamics of SynOV1.1 as well as type and severity of toxicity based on safety and tolerability assessments. Participants will receive administration bi weekly. 2 dose level will be evaluated based on part 1 result.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participates in the clinical trial study; fully understands the study and signs the ICF; and is willing to follow and will be able to complete all trial procedures.
2. Is ≥18 years old when signing ICF; male or female.
3. Has locally advanced or metastatic AFP-positive solid tumorsthat has relapsed or is refractory to standard cancer therapies, or where no standard therapies are available. AFP positive means that serum samples have levels of AFP> 20 ng/ml during screening or an AFP immunohistochemistry [IHC] test of previous tumor tissue samples was positive.
4. Has at least one lesion that cannot be surgically removed which can be injected directly or through ultrasound (US) and/or computer tomography (CT) guidance.
5. Has at least one measurable tumor lesion.
6. Has a Child-Pugh score of Class A.
7. Has an ECOG performance status is 0 to 1 one week prior to the treatment.
8. Has an expected survival time of ≥ 12 weeks.
9. Has limited alterations in hematology or clinical chemistry: ANC≥ 1.5 × 10^9/L, PLT≥ 75 × 109/L, TBIL≤ 1.5 ×ULN, AST and ALT≤5 × ULN, Alb≥ 2.8 g/dL, Crea≤ 1.5 × ULN, INR≤ 1.5 × ULN.
10. Agrees to provide archived or fresh tumor tissue specimens according to the individual's situation and blood samples.
11. A female participant who is postmenopausal, or whose serum pregnancy test result is negative. A woman who has not experienced a menstrual period for 12 months due to non-medical reasons is considered postmenopausal.
12. Female participants of child-bearing potential and male participants shall agree to take medically acceptable contraception measures (hormones, barrier, or abstinence) while on treatment and for 90 days following completion of treatment.

Exclusion Criteria:

1. Received any anti-tumor treatment within the 4 weeks prior to study drug administration. The anti-tumor treatment includes surgery, ethanol injection, radiofrequency ablation, trans-arterial chemoembolization, intrahepatic chemotherapy, chemotherapy, biotherapy, immunotherapy, hormone, or radiotherapy.
2. Received a systemic treatment of glucocorticoid (Prednisone > 10 mg/day or equivalent dose of a similar medicine) or other immunosuppressant treatment 14 days prior to study drug administration。
3. Administration of immune-regulating medicines within 14 days prior to study drug administration of the investigational drug。
4. Administration of live-attenuated vaccines within 4 weeks prior to study drug administration。
5. Previously treated with oncolytic viruses or other gene therapies.
6. Received treatment of unapproved investigational drugs within 4 weeks prior to study drug administration.
7. Currently participating in another clinical study, except for an observational or genetic (non-interventional) clinical study or a follow-up period.
8. Had major organ surgery (excluding biopsy) or had significant trauma within 4 weeks prior to study drug administration.
9. An adverse event from the previous anti-tumor therapy that has not resolved to ≤ Grade 1 or stabilized according to NCI-CTCAE v5.0, except for the adverse event of non-risk toxicity as judged by the investigator and sponsor.
10. Participants with clinical symptoms of central nervous system metastasis or meningeal metastasis, or other evidence demonstrating the central nervous system metastasis or meningeal metastasis has not been controlled.
11. History of meningococcal disease.
12. Evidence of uncontrolled severe comorbidity that may affect the participant's compliance with the study protocol, including severe liver disease (e.g. severe esophageal and gastric varices that require interventional treatment, cirrhosis, hepatic encephalopathy, or venous syndrome).
13. History of serious cardiovascular disease。
14. Participants who have third interstitial fluid beyond clinical control judged by the investigator.
15. History of tuberculosis infection or immunodeficiency, including participants who have tested positive for the human immunodeficiency virus (HIV) antibody.
16. Participants who are allergic to any component of the SynOV1.1 drug product.
17. Participants who are suffering from a known mental illness or substance abuse that may affect the objectivity of the trial.
18. Female participants who are pregnant, lactating, or who plan to get pregnant or to breastfeed during the trial.
19. Other reasons as judged by the investigator, including but not limited to highly vascularized tumors, exogenous, adjacent to necrotic areas, liver cysts, tumor site at the location with high risk of adverse events or not suitable for intratumoral injection, or tumor that will enhance the contraindications of CT/ MRI examination.
20. A significant bleeding event, as assessed by the investigator, that occurring within 12 months prior to study drug administration may increase the risk of intratumoral injection procedures.
21. Participants who cannot discontinue anticoagulant or antiplatelet medications prior to the intratumoral injection of SynOV1.1.
22. Participants who require treatment for active systemic infection.
23. Participants who have been diagnosed with bile duct cancer, bile duct liver cancer, fibrolamellar carcinoma, or hepatoblastoma based on histological finding.
24. Participants who have a severe inflammatory skin disease that currently requires medication or who have a history of severe eczema that requires medication.
25. Participants who received or plan to receive an organ transplant, such as a liver transplantation.
26. Participants who carry another type of tumor that has required active treatment in the past 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The dose-limiting toxicities (DLTs) of SynOV1.1 in patients with HCC | 30 months
  Incidence and nature of DLT of SynOV1.1 in in patients with HCC, graded according to NCI CTCAE v5
The maximum-tolerated dose (MTD) of SynOV1.1 in patients with HCC | 30 months
  MTD for patients with HCC received SynOV1.1 treatment.
The response rate of patients with HCC receiving SynOV1.1 | 30 months
  response rate based on RECIST ver. 1.1

SECONDARY OUTCOMES:
The biodistribution of SynOV1.1，as determined by the concentration of SynOV1.1 in blood of participating patients. | 30 months
  The concentration of SynOV1.1 in blood of participating patients will be measured by QT-PCR.
The immunogenicity of SynOV1.1, as determined by quantitation of neutralizing antibodies in blood of participating patients. | 30 months
  The quantitation of neutralizing antibodies in blood of participating patients will be measured by CPE.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 30 months
  Determine the number of participants who received SynOV1.1 in combination with Atezolizumab treatment with treatment-related adverse events, as assessed by the CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, MD, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China